CLINICAL TRIAL: NCT05097638
Title: Lung Health After Tuberculosis: Clinical and Functional Assessment in Post Pulmonary Tuberculosis Egyptian Patients.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen Aly Mahmoud Abdel Aleem, Lecture in Chest and Tuberculosis Department, Faculty of Medicine, Assiut University
Other Study IDs: 5884
Record Dates: First submitted 2021-10-07; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Tuberculoses; Pulmonary Function; Newborn, Abnormal
Keywords: pulmonary Tuberculosis; Spirometry; Pulmonary Function
MeSH Terms: conditions — Tuberculosis, Pulmonary; Antisocial Personality Disorder | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cured pulmonary Tuberculosis patients: 6 months after a completed course of anti-tuberculosis therapy
  Interventions: Diagnostic Test: spirometry

INTERVENTIONS:
Diagnostic Test: spirometry — Patient do spirometry

SUMMARY:
Some of pulmonary tuberculous patients who completed their medication course experience lung function impairment

DETAILED DESCRIPTION:
Some of pulmonary tuberculous patients who completed their medication course experience lung function impairment which may influence their quality of life. However, the pattern and nature of post-tuberculosis lung impairment is still not identified. Thus, the aim of this study was to determine the type and degree of lung physiology changes in previously treated tuberculous patients which latter may affect their quality of life; thus helping clinicians for early diagnosis of lung impairment, especially in tuberculous endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Patient completed an outpatient course of standard first line anti-tuberculosis therapy and declared as cured

Exclusion Criteria:

* Smoker (to avoid spirometry biases).
* Extrapulmonary tuberculosis cases
* Multidrug resistant tuberculosis
* known contraindications to spirometry testing
* Individuals with chest wall deformities or neuromuscular diseases
* Patients who failed to achieve acceptability and reproducibility criteria of the spirometry test
* Defaulter cases or irregular treatment,
* known coexisting chronic lung disease as history of asthma or interstitial lung diseases
* A history of illicit drug use
* Patients with comorbidities: renal and hepatic insufficiency, heart diseases and metabolic disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient more than 18 years old had been newly diagnosed drug-sensitive first episode pulmonary tuberculosis, confirmed by sputum smear microscopy were included in the study. He completed an outpatient course of standard first line anti-tuberculosis therapy (6 months) and declared as cured without radiological change over the past year (in comparable with chest X-ray at the end of TB treatment).
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Post tuberculosis lung functional impairment | 6 months
  spirometry abnormality either: restrictive, obstructive, or mixed
post tuberculosis persistent clinical symptoms | 6 months
  either cough , sputum , breathlessness, hemoptysis
Grading of obstruction function: | 6 months
  grading according to GOLD : mild , moderate , severe , very severe

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Department-faculty of medicine-Assuit university, Asyut, Egypt